CLINICAL TRIAL: NCT01441947
Title: A Phase II Trial of Cabozantinib in Women With Metastatic Hormone-Receptor-Positive Breast Cancer With Involvement of Bone
Brief Title: Cabozantinib in Women With Metastatic Hormone-Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Principal Investigator, Attending Physician in Medical Oncology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11-208
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: ER+; PR+; Human Epidermal Growth Factor Receptor (HER) 2 negative; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — cabozantinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Cabozantinib (Experimental): Oral cabozantinib therapy daily
  Interventions: Drug: Cabozantinib
- Cabozantinib plus fulvestrant (Experimental): Combination therapy with oral cabozantinib daily plus fulvestrant monthly Intramuscularly (IM)
  Interventions: Drug: Cabozantinib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Cabozantinib — Given orally daily with a starting dose of 40 mg
  Other Names: XL184
Drug: Fulvestrant — Given intramuscularly 500 mg on Days 1 and 15 of the first 28 day cycle, then on Day 1 only each cycle after
  Other Names: Faslodex
  Arms: Cabozantinib plus fulvestrant

SUMMARY:
The study drug cabozantinib works by inhibiting several different proteins which are believed to be involved in breast cancer tumor growth, its ability to spread, and its ability to form new blood vessels. This drug has been used in other research studies and information from those other research studies suggests that this drug may help to prevent cancer growth.

The single agent portion of this study is now closed to accrual. This research study is now examining the efficacy of cabozantinib in combination with fulvestrant for treatment of hormone-receptor-positive breast cancer that has spread to bone.

DETAILED DESCRIPTION:
Cabozantinib will be taken orally once a day in cycles of 28 days (4 weeks). Fulvestrant will be given intramuscularly on days 1 and 15 of cycle 1 and on day 1 of all subsequent cycles.

On Day 1 of each cycle subjects will have the following tests and procedures:

* Performance status
* Physical exam
* Vital signs
* Routine blood samples
* Blood and urine samples to look at bone markers (Cycle 1 through 6 only)

Subjects will also have the following additional tests and procedures:

* Tumor assessment by Computed Tomography (CT) scan and bone scan at Cycle 3, then every 12 weeks
* Blood or urine pregnancy test (if applicable) on Day 1 of Cycles 1, 2, 4, then every 12 weeks
* Urine sample and blood test for thyroid function (Cycle 1, 3, 5, then every 6 weeks)
* Blood test for breast cancer tumor marker (Cycle 1 and 4, then every 6 weeks)
* Pain questionnaire and painkiller medication diary at 7-day intervals during Week 3, Week 6, and every 6 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Clear evidence of metastases to bone on isotope bone scan
* Histologically or cytologically confirmed metastatic Estrogen-receptor-positive (ER+) and/or Progesterone-receptor-positive (PR+) and Human Epidermal Growth Factor Receptor (HER) 2 negative breast cancer
* Received at least one prior line of hormonal or chemo-therapy for metastatic disease
* must be post menopausal
* Recovered from toxicities related to prior treatment, except alopecia, lymphopenia, or other non-clinically significant Adverse Events (AEs)
* Life expectancy > 3 months
* Adequate organ and marrow function
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception
* Able to lie flat for up to 45 minutes for imaging studies
* Able to swallow capsules or tablets

Exclusion Criteria:

* Pregnant or breast-feeding
* Has experienced clinically-significant hematemesis or hemoptysis of > 0.5 teaspoons of red blood, or other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* Untreated, symptomatic or uncontrolled brain metastasis requiring current treatment including steroids and anti-convulsants
* more than 1 prior line of chemotherapy for treatment of metastatic breast cancer
* prior treatment with fulvestrant
* Requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or coumadin-related agents, thrombin or Factor Xa inhibitors, and antiplatelet agents (eg, clopidogrel)
* Uncontrolled or significant intercurrent illness
* Gastrointestinal disorders, particularly those associated with a high risk of perforation or fistula formation
* Active infection requiring systemic treatment
* Serious non-healing wound/ulcer/bone fracture
* History of organ transplant
* Concurrent uncompensated hypothyroidism or thyroid dysfunction
* Previously-identified allergy or hypersensitivity to components of the study treatment formulation
* Diagnosis of another malignancy, requiring systemic treatment, within the last 2 years, unless non-melanoma skin cancer, in-situ carcinoma of the cervix, or superficial bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Isakoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Higgins MJ, Tolaney SM, Come SE, Smith MR, Fornier M, Mahmood U, Baselga J, Yeap BY, Chabner BA, Isakoff SJ. A Phase II Trial of Cabozantinib in Hormone Receptor-Positive Breast Cancer with Bone Metastases. Oncologist. 2020 Aug;25(8):652-660. doi: 10.1634/theoncologist.2020-0127. Epub 2020 Jun 18. PMID 32463152

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib | Cabozantinib Plus Fulvestrant
Started | 55 | 13
Completed | 52 | 13
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib | Cabozantinib Plus Fulvestrant | Total
Number analyzed (Participants) | 55 | 13 | 68
Age, Continuous [Median (Full Range); unit: years] | 55 [33 to 79] | 63 [51 to 78] | 56 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 13 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 12 | 56
  Unknown or Not Reported | 11 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 45 | 12 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Bone Scan Response Rate
Description: Bone scan response rate will be defined as the percentage of patients experiencing a complete resolution of bone lesions or partial response in the isotope bone scan per Bone Scan Time Point Response Criteria, as defined in the protocol. Complete resolution is defined as the disappearance of all areas of radiotracer uptake attributable to metastatic disease, and a partial response is defined as significant improvement in radiotracer uptake in areas attributable to metastatic disease, but not meeting the criteria for CR.
Time Frame: 2 years
Population: 55 patients initially enrolled to the Cabozantinib cohort, but 3 withdrew prior to starting study treatment. Per protocol section 14.1, only patients in the main cabozantinib cohort were included in the primary analysis. There are no primary endpoints for the pilot cabozantinib/ fulvestrant cohort.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 52
percentage of participants | 38.5 [27.1 to 51.0]

2. Secondary Outcome: Overall Response Rate by RECIST v 1.1
Description: The overall response rate (ORR) is defined as the percentage of patients experiencing a complete response or partial response on PET imaging per mRECIST (modified response evaluation criteria in solid tumors), as defined in the protocol. A complete response is defined as resolution of all areas of FDG uptake attributable to metastatic disease. A partial response is defined as significantly decreased FDG uptake in areas attributable to metastatic disease, but not meeting the criteria for a complete response.
Time Frame: 2 years
Population: 55 patients initially enrolled to the Cabozantinib cohort, but 3 withdrew prior to starting study treatment. Per protocol section 14.4, ORR is a secondary endpoint only for the main cabozantinib cohort; endpoints for the pilot cohort are listed separately. Additionally, per protocol section 14.4, "All secondary endpoint analyses of this trial are considered exploratory." Results for ORR are available, so we are reporting them here even though this endpoint was considered exploratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 52
Participants | 0

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the difference between the date of a patient's enrollment onto this study until the date of death. Patients who are alive at last contact will be censored for OS at this date.
Time Frame: 5 years
Population: 55 patients initially enrolled to the Cabozantinib cohort, but 3 withdrew prior to starting study treatment. Per protocol section 14.4, OS is a secondary endpoint only for the main cabozantinib cohort; endpoints for the pilot cohort are listed separately. Additionally, per protocol section 14.4, "All secondary endpoint analyses of this trial are considered exploratory." Results for OS are available, so we are reporting them here even though this endpoint was considered exploratory.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 52
months | 19.6 [18.0 to 26.8]

4. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the difference between the date of a patient's enrollment onto this study until the earlier of the date of progression or the date of death. Patients who are alive and progression-free at last contact will be censored for PFS at this date.
Time Frame: 5 years
Population: 55 patients initially enrolled to the Cabozantinib cohort, but 3 withdrew prior to starting study treatment. Per protocol section 14.4, PFS is a secondary endpoint only for the main cabozantinib cohort; endpoints for the pilot cohort are listed separately. Additionally, per protocol section 14.4, "All secondary endpoint analyses of this trial are considered exploratory." Results for PFS are available, so we are reporting them here even though this endpoint was considered exploratory.
Measure: Median (90% Confidence Interval); unit: units on a scale
Arm/Group | Cabozantinib
Number analyzed (Participants) | 52
units on a scale | 4.3 [2.8 to 5.5]

ADVERSE EVENTS:
Time Frame: Adverse event reporting will begin from the time of the first dose of study treatment, through the study and until the final study visit (up to 5 years)
Arm/Group | Cabozantinib | Cabozantinib Plus Fulvestrant
All-Cause Mortality (participants affected / at risk) | 35/52 | 12/13
Serious Adverse Events (participants affected / at risk) | 13/52 | 3/13
Other Adverse Events (participants affected / at risk) | 51/52 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=52) | Cabozantinib Plus Fulvestrant (N=13)
Pathologic left femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Vulval Infection (Infections and infestations) | 1 | 0
Concentration Impairment (Nervous system disorders) | 1 | 0
Fractured C7, T5 (Injury, poisoning and procedural complications) | 1 | 0
Death (General disorders) | 3 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute Interstitial Nephritis (Renal and urinary disorders) | 1 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Impending pathologic fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Decrease in LVEF (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Respiratory Failure (Infections and infestations) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilateral pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vascular access complication (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=52) | Cabozantinib Plus Fulvestrant (N=13)
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Activated partial thromboplastin time prolonged (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 28 | 5
Alkaline phosphatase increased (Investigations) | 19 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3
Anemia (Blood and lymphatic system disorders) | 6 | 2
Anorexia (Metabolism and nutrition disorders) | 19 | 8
Anxiety (Psychiatric disorders) | 1 | 1
Aphonia (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 28 | 5
Ataxia (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 3
Bloating (Gastrointestinal disorders) | 1 | 2
Blood and lymphatic system disorders - Other, specify: decreased hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify: decreased potassium (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 5 | 0
Blurred vision (Eye disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 3
Breast pain (Reproductive system and breast disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac disorders - Other, specify: cardiac arrhythmia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0
Chills (General disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depression (Psychiatric disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 26 | 6
Dizziness (Nervous system disorders) | 5 | 0
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0
Dysesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 10 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Ear and labyrinth disorders - Other, specify: ear block (Ear and labyrinth disorders) | 1 | 0
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 4
Endocrine disorders - Other, specify: TSH elevation (Endocrine disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 | 0
Esophagitis (Gastrointestinal disorders) | 5 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Eye disorders - Other, specify: change in iris color (Eye disorders) | 1 | 0
Eye disorders - Other, specify: Diplopia (Eye disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fat atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 37 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Fever (General disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 4 | 3
Flushing (Vascular disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 3 | 0
Gait disturbance (General disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 5
Gastrointestinal disorders - Other, specify: Oral petichiae/papules (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: heart burn (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: taste alteration (Gastrointestinal disorders) | 8 | 0
Gastrointestinal disorders - Other, specify: reflux (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: Tongue soreness (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: loose stool (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other, specify: hair turning grey (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify: oral thrush (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify: jaw numbness (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
General disorders and administration site conditions - Other, specify: feet sensitivities (General disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gum infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 13 | 4
Hemoglobin increased (Investigations) | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Hepatobiliary disorders - Other, specify: LDH elevation (Hepatobiliary disorders) | 7 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Hot flashes (Vascular disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hypertension (Vascular disorders) | 17 | 3
Hyperthyroidism (Endocrine disorders) | 4 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 8 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 8 | 1
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 13 | 2
Hypothyroidism (Endocrine disorders) | 12 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Investigations - Other, specify: Decreased hemoglobin (Investigations) | 2 | 0
Investigations - Other, specify: TSH elevation (Investigations) | 5 | 0
Investigations - Other, specify: total protein decreased (Investigations) | 3 | 0
Investigations - Other, specify (Investigations) | 2 | 0
Investigations - Other, specify: thrombocytosis (Investigations) | 2 | 0
Investigations - Other, specify: Urine Protein Creatinine Ratio - present at baseline (Investigations) | 1 | 0
Investigations - Other, specify: blood urea nitrogen increased (Investigations) | 1 | 0
Investigations - Other, specify: amylase increased (Investigations) | 1 | 0
Investigations - Other, specify: white blood cells in urine (Investigations) | 0 | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lipase increased (Investigations) | 7 | 3
Lung infection (Infections and infestations) | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 12 | 0
Mediastinal infection (Infections and infestations) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Metabolism and nutrition disorders - Other, specify: hypochloridemia (Metabolism and nutrition disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 19 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify: leg cramping (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal and connective tissue disorder - Other, specify: achiness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: left leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: right rib pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: hand cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: bilateral leg heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify: pleuritic pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 24 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Nervous system disorders - Other, specify: dysphonia (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: neuropathy in fingers (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: intermittent lightheadedness (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: right leg nerve pain (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 5 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 3 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain (General disorders) | 17 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 | 3
Palpitations (Cardiac disorders) | 2 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 0
Phlebitis (Vascular disorders) | 0 | 1
Platelet count decreased (Investigations) | 6 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify: pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 0
Salivary gland infection (Infections and infestations) | 1 | 0
Serum amylase increased (Investigations) | 5 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: skin rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: hair thinning (Skin and subcutaneous tissue disorders) | 5 | 0
Skin and subcutaneous tissue disorders - Other, specify: hair depigmentation (Skin and subcutaneous tissue disorders) | 7 | 0
Skin and subcutaneous tissue disorders - Other, specify: skin peeling bilateral soles of feet (Skin and subcutaneous tissue disorders) | 1 | 0 — possible verrucous infection
Skin and subcutaneous tissue disorders - Other, specify: acne vulgaris (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: tick bite (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: hair discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: right great toe ingrown toenail (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify: wart (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: rash on scalp (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: rash on arms (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify: tender soles of feet (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Skin/subcutaneous tissue disorders; Other, specify: PPE (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Spasticity (Nervous system disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Tooth infection (Infections and infestations) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 10 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 15 | 4
White blood cell decreased (Investigations) | 18 | 1

LIMITATIONS AND CAVEATS:
Primary (bone scan response rate) and reported secondary (ORR, OS, PFS) objectives are only applicable for the main cohort (Cabozantinib only), and objectives for the pilot cohort are listed separately. Per protocol section 14, "all secondary endpoint analyses of this trial are considered exploratory." We reported the secondary objectives for the main cohort listed above despite these being considered exploratory, as they were readily available. The remaining exploratory analyses were not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT01441947/Prot_SAP_000.pdf